CLINICAL TRIAL: NCT04146259
Title: Changes in Circulating Sclerostin Levels During Acute Postsurgical Hypoparathyroidism
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Symeon tournis, Senior Research Fellow, University of Athens
Other Study IDs: 1387/08-12-2015
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Hypoparathyroidism Postprocedural
Keywords: Sclerostin; Hypoparathyroidism
MeSH Terms: conditions — Sclerosteosis; Hypoparathyroidism | interventions — Calcium Carbonate; alfacalcidol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: Control
- Group B: Post-surgical hypoparathyroidism
  Interventions: Drug: calcium carbonate and alphacalcidol

INTERVENTIONS:
Drug: calcium carbonate and alphacalcidol — treatment for hypocalcemia
  Groups: Group B

SUMMARY:
To investigate changes in sclerostin levels following acute post-thyroidectomy hypoparathyroidism

DETAILED DESCRIPTION:
Female patients with thyroid disorders, referred to the Department of Head and Neck Surgery, at Metaxa Anti-Cancer Hospital of Piraeus, for total thyroidectomy.

Based on the development of biochemical hypocalcemia (cCa < 8.4 mg/dl), subjects were divided into 2 groups: Group A: without postsurgical hypoparathyroidism that served as controls and group B: subjects, with acute postsurgical hypoparathyroidism.

Blood collections were performed in the morning after an overnight fast, in at least 3 different time points; preoperatively, 1st postoperative day and 7th postoperative day for the detrmination of sclerostin levels

ELIGIBILITY:
Inclusion Criteria:

* Indication for total thyroidectomy

Exclusion Criteria:

* parathyroid disorders, chronic kidney disease (eGFR< 60 ml/min), treatment with antiosteoporosis drugs, rheumatic disease and history of long term (>1 month) or current corticosteroid use

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female patients with indication for total thyroidectomy
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
change in circulating serum sclerostin levels (pmol/L) during the observation period | 7 days
  change in circulating serum sclerostin levels (pmol/L)during the observation period

SECONDARY OUTCOMES:
the between groups difference in % changes of circulating sclerostin | 7 days
  the between groups difference in % changes of circulating sclerostin

CONTACTS AND LOCATIONS:
Locations (1):
- Symeon Tournis, Athens, Greece

IPD SHARING:
Plan to Share IPD: No